CLINICAL TRIAL: NCT01038830
Title: The Change in Level of Interferon-gamma Assay in Active Tuberculosis Patients During Treatment
Brief Title: QuantiFERON Change During Anti-tuberculosis Medication
Status: Completed | Type: Observational
Sponsor: Armed Forces Capital Hospital, Republic of Korea (Other Government)
Responsible Party: Sei Won Lee/Division chief of pulmonology, Armed Forces Capital Hospital
Other Study IDs: QFTchange
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2009-12

CONDITIONS: Tuberculosis; Interferon-gamma Release Assay
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the change of QuantiFERON-TB gold in tube assay (QFT) during the treatment of active tuberculosis.

DETAILED DESCRIPTION:
Patients with active pulmonary tuberculosis are enrolled and, QFTs are performed for each subjects before treatment and 1, 3, 6 months after treatment. Investigators check the level of interferon-gamma, and reversion and conversion of this test.

ELIGIBILITY:
Inclusion Criteria:

* All subjects with active tuberculosis

Exclusion Criteria:

* Subjects who cannot complete study
* Subjects who have taken anti-tuberculosis medication for more than a month before visit of our hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Young healthy subjects in Korean military
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Capital Hospital, Seongnam-si, Gyeonggi-do, South Korea